CLINICAL TRIAL: NCT04339270
Title: Chronic Airway Disease, Mucus Rheology and Exacerbations: a Randomized Controlled Trial of COPD Patients
Brief Title: Chronic Airway Disease, Mucus Rheology and Exacerbations
Acronym: COPD-CARhE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Rheonova (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RECHMPL19_0074
Record Dates: First submitted 2020-04-02; First posted 2020-04-09 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial comparing outcomes in 2 parallel arms (36 vs 36 patients).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: CASA-Q scoring is performed by the patient and then sealed away from investigator-view. Similarly, mucus rheology results are blinded. The patient does not know what arm he/she is in, as so does not know exactly why the prescription was made or not.
  Similarly, investigators/outcome assessors are blinded to both CASA-Q scores and sputum rheology. The prescription strategy is determined according to an algorithm, and investigators/outcome assessors do not know what arm the patient is in nor exactly why a prescription was made or not.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Azithromycin according to symptoms (Active Comparator): Patients randomized to this arm will be prescribed azithromycin in function of their symptoms.
  Interventions: Drug: Azithropycin according to symptoms
- Azithromycin according to rheology (Experimental): Patients randomized to this arm will be prescribed azithromycin in function of their sputum rheology.
  Interventions: Drug: Azithromycin according to rheology or symptoms

INTERVENTIONS:
Drug: Azithropycin according to symptoms — Patients randomized to the "standardized comparator arm" will benefit from the standard treatment for COPD, including with regard to the prescription of azithromycin in case of severe sputum complaints (here defined by a CASA-Q sputum symptoms score <70 to homogenize practices between centers).
  CASA-Q will be evaluated every 3 months.
  * If the patient has a sputum symptoms score <70, a prescription for 3 months of azithromycin treatment will be initiated. This prescription can be renewed every 3 months during the 12 months of follow-up planned in this study, if the patient continues to obtain a sputum symptoms score <70.
  * If the patient has a sputum symptoms score> 70, management is not changed.
  Arms: Azithromycin according to symptoms
Drug: Azithromycin according to rheology or symptoms — Treatment according to standard COPD management, except for the prescription of azithromycin, which will be prescribed in function of mucus rheology or as a function of sputum complaints (here defined by a CASA-Q sputum symptoms score <70).
  The rheology of mucus will be quantified every 3 months.
  * If the patient has spontaneous or induced sputum, and this sputum has a critical constraint (tau-C) > 39, a prescription for 3 months of azithromycin treatment will be initiated. This prescription may be renewed every 3 months during the 12 months of follow-up planned in this study.
  * If the patient has a sputum symptoms score <70, a prescription for 3 months of azithromycin treatment will be initiated. This prescription can be renewed every 3 months during the 12 months of follow-up planned in this study, if the patient continues to obtain a sputum symptoms score <70.
  * If the patient has a sputum symptoms score> 70, management is not changed.
  Arms: Azithromycin according to rheology

SUMMARY:
The main objective of this trial is to compare the exacerbation number over 12 months of follow-up between a group of patients with COPD treated according to standardized management (azithromycin prescribed in the event of severe sputum according to the CASA-Q score , standardized comparator arm) and a similar group in which azithromycin is prescribed based on mucus rheology (experimental arm) or CASA-Q.

DETAILED DESCRIPTION:
The secondary objectives are to compare between the 2 arms:

* exacerbation number according to their severity (observed throughout the duration of the study);
* the evolution of the symptoms, the rheology of the sputum, and the pulmonary function (measurements repeated every three months);
* medication consumption and adverse events (monitored throughout the duration of the study);
* patient trajectories during follow-up;
* the overall clinical improvement at the end of the study and the evolution of the quality of life (measurements repeated every 3 months);
* the change in biomarkers of interest (baseline versus end of study).

ELIGIBILITY:
Inclusion Criteria:

* Subjets between 40 - 85 years (included)
* Written and signed informed consent form
* Subjects must be able to attend all planned visits and comply with all test procedures
* Beneficiary of or affiliated with the French social security system
* Man or woman with chronic obstructive pulmonary disease for at least 1 year defined according to Global Initiative for Chronic Obstructive Lung Disease (GOLD) criteria and validated by the clinical investigator
* Optimal treatment according to GOLD class severity C or D recommendations
* >=3 exacerbation (regardless of severity: mild-moderate-severe) or ≥ 1 severe exacerbations (requiring hospitalization) in the past 12 months
* Spontaneous or induced sputum production
* Electrocardiogram: corrected distance between Q and T waves (QTC) <450 ms in men, QTC <470 ms in women
* Normal audiogram for age or absence of contraindication to azithromycin for long course according to Oto-Rhino-Laryngological specialist opinion

Exclusion Criteria:

* Pregnancy or breastfeeding
* Patients who are prisoners or under other forms of judicial protection
* Patients under any form of guardianship
* Participation in another interventional protocol, (current or during the month preceding inclusion)
* Received azithromycin in the past 3 months
* Patient whose primary diagnosis is bronchial dilation based on CT scan documentation
* Known hypersensitivity to azithromycin, erythromycin, any other macrolide, ketolide or any of the excipients of the azithromycin-based specialty used
* Concomitant use of medication contraindicated with azithromycin (dihydroergotamine, ergotamine, cisapride, colchicine)
* Other respiratory diseases or associated lung infections
* Severe hepatic insufficiency and severe cholestasis (a liver biological test will be carried out if clinical suspicion)
* Renal impairment with creatinine clearance < 40 mL/min
* Patients with hematological malignancies who have undergone allogeneic hematopoietic stem cell transplantation
* Patients with galactose intolerance, Lapp lactase deficiency or glucose or galactose malabsorption syndrome (rare hereditary disease) due to the presence of lactose in the specialty Zithromax.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-02-03 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
The main outcome measure is the number of exacerbations over the 12 months of follow-up. | 12 months
  An exacerbation is defined according to French recommendations as an "acute event characterized by worsening of respiratory symptoms (notably cough, sputum and dyspnea) beyond [normal] daily variation and leading to a modification of treatment: either a simple increase in bronchodilators (in this case, a duration greater than 24 hours is required to define an exacerbation) or the addition of another treatment (antibiotic therapy and / or oral corticosteroid therapy)."

SECONDARY OUTCOMES:
The number of mild exacerbations throughout follow-up | 12 months
  A mild exacerbation does not require new additional medicine.
The number of moderate exacerbations throughout follow-up | 12 months
  Moderate exacerbations require antibiotics or oral corticosteroids (but not hospitalization).
The number of severe exacerbations throughout follow-up | 12 months
  Severe exacerbations require hospitalization.
COPD Assessment Test (CAT) | Baseline (Day 0)
  Scores range from 0-40 with higher scores indicative of greater COPD impact on health status.
COPD Assessment Test (CAT) | 3 months
  Scores range from 0-40 with higher scores indicative of greater COPD impact on health status.
COPD Assessment Test (CAT) | 6 months
  Scores range from 0-40 with higher scores indicative of greater COPD impact on health status.
COPD Assessment Test (CAT) | 9 months
  Scores range from 0-40 with higher scores indicative of greater COPD impact on health status.
COPD Assessment Test (CAT) | 12 months
  Scores range from 0-40 with higher scores indicative of greater COPD impact on health status.
Sino Nasal Outcome Test 22 | Baseline (Day 0)
  The 22-question SNOT-22 is scored as 0 (no problem) to 5 (problem as bad as it can be) with a total range from 0 to 110 (higher scores indicate poorer outcomes).
Sino Nasal Outcome Test 22 | 3 months
  The 22-question SNOT-22 is scored as 0 (no problem) to 5 (problem as bad as it can be) with a total range from 0 to 110 (higher scores indicate poorer outcomes).
Sino Nasal Outcome Test 22 | 6 months
  The 22-question SNOT-22 is scored as 0 (no problem) to 5 (problem as bad as it can be) with a total range from 0 to 110 (higher scores indicate poorer outcomes).
Sino Nasal Outcome Test 22 | 9 months
  The 22-question SNOT-22 is scored as 0 (no problem) to 5 (problem as bad as it can be) with a total range from 0 to 110 (higher scores indicate poorer outcomes).
Sino Nasal Outcome Test 22 | 12 months
  The 22-question SNOT-22 is scored as 0 (no problem) to 5 (problem as bad as it can be) with a total range from 0 to 110 (higher scores indicate poorer outcomes).
Cough and sputum assessment questionnaire (CASA-Q) | Baseline (Day 0)
  The four domains of the CASA-Q (cough/sputum symptom and impact) use scales from 0 to 100, with lower scores indicating higher symptom/impact levels. The 20-item questionnaire with a 7-day recall assesses the frequency and severity of cough and sputum and their impact on everyday life in clinical (trial) settings.
Cough and sputum assessment questionnaire (CASA-Q) | 3 months
  The four domains of the CASA-Q (cough/sputum symptom and impact) use scales from 0 to 100, with lower scores indicating higher symptom/impact levels. The 20-item questionnaire with a 7-day recall assesses the frequency and severity of cough and sputum and their impact on everyday life in clinical (trial) settings.
Cough and sputum assessment questionnaire (CASA-Q) | 6 months
  The four domains of the CASA-Q (cough/sputum symptom and impact) use scales from 0 to 100, with lower scores indicating higher symptom/impact levels. The 20-item questionnaire with a 7-day recall assesses the frequency and severity of cough and sputum and their impact on everyday life in clinical (trial) settings.
Cough and sputum assessment questionnaire (CASA-Q) | 9 months
  The four domains of the CASA-Q (cough/sputum symptom and impact) use scales from 0 to 100, with lower scores indicating higher symptom/impact levels. The 20-item questionnaire with a 7-day recall assesses the frequency and severity of cough and sputum and their impact on everyday life in clinical (trial) settings.
Cough and sputum assessment questionnaire (CASA-Q) | 12 months
  The four domains of the CASA-Q (cough/sputum symptom and impact) use scales from 0 to 100, with lower scores indicating higher symptom/impact levels. The 20-item questionnaire with a 7-day recall assesses the frequency and severity of cough and sputum and their impact on everyday life in clinical (trial) settings.
Visual analogue scale for dyspnea | Baseline (Day 0)
  A patient-reported visual analogue scale (VAS) starting at 0 (no symptoms) and ending at 100 (the worst possible level of dyspnea possible).
Visual analogue scale for dyspnea | 3 months
  A patient-reported visual analogue scale (VAS) starting at 0 (no symptoms) and ending at 100 (the worst possible level of dyspnea possible).
Visual analogue scale for dyspnea | 6 months
  A patient-reported visual analogue scale (VAS) starting at 0 (no symptoms) and ending at 100 (the worst possible level of dyspnea possible).
Visual analogue scale for dyspnea | 9 months
  A patient-reported visual analogue scale (VAS) starting at 0 (no symptoms) and ending at 100 (the worst possible level of dyspnea possible).
Visual analogue scale for dyspnea | 12 months
  A patient-reported visual analogue scale (VAS) starting at 0 (no symptoms) and ending at 100 (the worst possible level of dyspnea possible).
Visual analogue scale for coughing | Baseline (Day 0)
  A patient-reported visual analogue scale (VAS) starting at 0 (no symptoms) and ending at 100 (the worst possible level of coughing possible).
Visual analogue scale for coughing | 3 months
  A patient-reported visual analogue scale (VAS) starting at 0 (no symptoms) and ending at 100 (the worst possible level of coughing possible).
Visual analogue scale for coughing | 6 months
  A patient-reported visual analogue scale (VAS) starting at 0 (no symptoms) and ending at 100 (the worst possible level of coughing possible).
Visual analogue scale for coughing | 9 months
  A patient-reported visual analogue scale (VAS) starting at 0 (no symptoms) and ending at 100 (the worst possible level of coughing possible).
Visual analogue scale for coughing | 12 months
  A patient-reported visual analogue scale (VAS) starting at 0 (no symptoms) and ending at 100 (the worst possible level of coughing possible).
Visual analogue scale for sputum production | Baseline (Day 0)
  A patient-reported visual analogue scale (VAS) starting at 0 (no symptoms) and ending at 100 (the worst possible level of sputum production possible).
Visual analogue scale for sputum production | 3 months
  A patient-reported visual analogue scale (VAS) starting at 0 (no symptoms) and ending at 100 (the worst possible level of sputum production possible).
Visual analogue scale for sputum production | 6 months
  A patient-reported visual analogue scale (VAS) starting at 0 (no symptoms) and ending at 100 (the worst possible level of sputum production possible).
Visual analogue scale for sputum production | 9 months
  A patient-reported visual analogue scale (VAS) starting at 0 (no symptoms) and ending at 100 (the worst possible level of sputum production possible).
Visual analogue scale for sputum production | 12 months
  A patient-reported visual analogue scale (VAS) starting at 0 (no symptoms) and ending at 100 (the worst possible level of sputum production possible).
Rheology: modulus of elasticity of mucus (G ') | Baseline (Day 0)
Rheology: modulus of elasticity of mucus (G ') | 3 months
Rheology: modulus of elasticity of mucus (G ') | 6 months
Rheology: modulus of elasticity of mucus (G ') | 9 months
Rheology: modulus of elasticity of mucus (G ') | 12 months
Rheology: the viscous module (G '') | Baseline (Day 0)
Rheology: the viscous module (G '') | 3 months
Rheology: the viscous module (G '') | 6 months
Rheology: the viscous module (G '') | 9 months
Rheology: the viscous module (G '') | 12 months
Rheology: The ratio G '' / G ' | Baseline (Day 0)
Rheology: The ratio G '' / G ' | 3 months
Rheology: The ratio G '' / G ' | 6 months
Rheology: The ratio G '' / G ' | 9 months
Rheology: The ratio G '' / G ' | 12 months
Rheology: the critical constraint (tau-C). | Baseline (Day 0)
Rheology: the critical constraint (tau-C). | 3 months
Rheology: the critical constraint (tau-C). | 6 months
Rheology: the critical constraint (tau-C). | 9 months
Rheology: the critical constraint (tau-C). | 12 months
Spirometry: forced expiratory volume in 1 minute (FEV1) | Baseline (day 0)
Spirometry: forced expiratory volume in 1 minute (FEV1) | 3 months
Spirometry: forced expiratory volume in 1 minute (FEV1) | 6 months
Spirometry: forced expiratory volume in 1 minute (FEV1) | 9 months
Spirometry: forced expiratory volume in 1 minute (FEV1) | 12 months
Spirometry: forced vital capacity (FVC) | Baseline (day 0)
Spirometry: forced vital capacity (FVC) | 3 months
Spirometry: forced vital capacity (FVC) | 6 months
Spirometry: forced vital capacity (FVC) | 9 months
Spirometry: forced vital capacity (FVC) | 12 months
Spirometry: FEV1/FVC | Baseline (day 0)
Spirometry: FEV1/FVC | 3 months
Spirometry: FEV1/FVC | 6 months
Spirometry: FEV1/FVC | 9 months
Spirometry: FEV1/FVC | 12 months
Plethysmography for lung volumes: residual volume (RV) | Baseline (day 0)
Plethysmography for lung volumes: residual volume (RV) | 3 months
Plethysmography for lung volumes: residual volume (RV) | 6 months
Plethysmography for lung volumes: residual volume (RV) | 9 months
Plethysmography for lung volumes: residual volume (RV) | 12 months
Plethysmography for lung volumes: functional residual capacity (FRC) | Baseline (day 0)
Plethysmography for lung volumes: functional residual capacity (FRC) | 3 months
Plethysmography for lung volumes: functional residual capacity (FRC) | 6 months
Plethysmography for lung volumes: functional residual capacity (FRC) | 9 months
Plethysmography for lung volumes: functional residual capacity (FRC) | 12 months
Plethysmography for lung volumes: total lung capacity (TLC) | Baseline (day 0)
Plethysmography for lung volumes: total lung capacity (TLC) | 3 months
Plethysmography for lung volumes: total lung capacity (TLC) | 6 months
Plethysmography for lung volumes: total lung capacity (TLC) | 9 months
Plethysmography for lung volumes: total lung capacity (TLC) | 12 months
Plethysmography for lung volumes: RV/TLC | Baseline (day 0)
Plethysmography for lung volumes: RV/TLC | 3 months
Plethysmography for lung volumes: RV/TLC | 6 months
Plethysmography for lung volumes: RV/TLC | 9 months
Plethysmography for lung volumes: RV/TLC | 12 months
Drug consumption throughout the study. | 12 months
The number of adverse events will be recorded throughout the study. | 12 months
Episodes of exacerbation throughout the study | 12 months
  For each exacerbation, the beginning and end dates will be recorded.
Episodes of hospitalization throughout the study | 12 months
  For each hospitalization, the beginning and end dates will be recorded.
Clinical improvement | 12 months
  Clinical improvement is scored via a point system from 0 to 3 at the end of the study. The points are added-up as follows:
  * 1 point: no more than one exacerbation without hospitalization during the 52 weeks of follow-up;
  * 1 point: gain > 100mL in pre-bronchodilator FEV1 at the 52nd week compared to the baseline state;
  * 1 point: variation of the CAT score during the 52 weeks of observation > 2.
Medical outcomes study 36-Item Short Form Survey (SF-36) | Baseline (day 0)
  The SF-36 taps eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. It also includes a single item that provides an indication of perceived change in health. A score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Medical outcomes study 36-Item Short Form Survey (SF-36) | 3 months
  The SF-36 taps eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. It also includes a single item that provides an indication of perceived change in health. A score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Medical outcomes study 36-Item Short Form Survey (SF-36) | 6 months
  The SF-36 taps eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. It also includes a single item that provides an indication of perceived change in health. A score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Medical outcomes study 36-Item Short Form Survey (SF-36) | 9 months
  The SF-36 taps eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. It also includes a single item that provides an indication of perceived change in health. A score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Medical outcomes study 36-Item Short Form Survey (SF-36) | 12 months
  The SF-36 taps eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. It also includes a single item that provides an indication of perceived change in health. A score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
EQ-5D-5L | Baseline (day 0)
  In its original version, this self-administered questionnaire consists of two pages: the first contains the EQ-5D descriptive system and the second a visual analogue scale. The descriptive system has five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), each described by five levels of intensity ("no problems", "slight problems", "moderate problems", "severe problems" and "extreme problems or complete inability"). The respondent must indicate one intensity level for each dimension.
EQ-5D-5L | 3 months
  In its original version, this self-administered questionnaire consists of two pages: the first contains the EQ-5D descriptive system and the second a visual analogue scale. The descriptive system has five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), each described by five levels of intensity ("no problems", "slight problems", "moderate problems", "severe problems" and "extreme problems or complete inability"). The respondent must indicate one intensity level for each dimension.
EQ-5D-5L | 6 months
  In its original version, this self-administered questionnaire consists of two pages: the first contains the EQ-5D descriptive system and the second a visual analogue scale. The descriptive system has five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), each described by five levels of intensity ("no problems", "slight problems", "moderate problems", "severe problems" and "extreme problems or complete inability"). The respondent must indicate one intensity level for each dimension.
EQ-5D-5L | 9 months
  In its original version, this self-administered questionnaire consists of two pages: the first contains the EQ-5D descriptive system and the second a visual analogue scale. The descriptive system has five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), each described by five levels of intensity ("no problems", "slight problems", "moderate problems", "severe problems" and "extreme problems or complete inability"). The respondent must indicate one intensity level for each dimension.
EQ-5D-5L | 12 months
  In its original version, this self-administered questionnaire consists of two pages: the first contains the EQ-5D descriptive system and the second a visual analogue scale. The descriptive system has five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), each described by five levels of intensity ("no problems", "slight problems", "moderate problems", "severe problems" and "extreme problems or complete inability"). The respondent must indicate one intensity level for each dimension.
St-George's Respiratory Questionnaire | Baseline (day 0)
  Scores range from 0 to 100, with higher scores indicating more limitations.
St-George's Respiratory Questionnaire | 3 months
  Scores range from 0 to 100, with higher scores indicating more limitations.
St-George's Respiratory Questionnaire | 6 months
  Scores range from 0 to 100, with higher scores indicating more limitations.
St-George's Respiratory Questionnaire | 9 months
  Scores range from 0 to 100, with higher scores indicating more limitations.
St-George's Respiratory Questionnaire | 12 months
  Scores range from 0 to 100, with higher scores indicating more limitations.
Blood cell differential: neutrophil levels | Baseline (day 0)
  A complete blood cell differential will be taken, including neutrophilia and eosinophilia.
Blood cell differential: eosinophil levels | Baseline (day 0)
  A complete blood cell differential will be taken, including neutrophilia and eosinophilia.
Blood cell differential: neutrophil levels | 12 months
  A complete blood cell differential will be taken, including neutrophilia and eosinophilia.
Blood cell differential: eosinophil levels | 12 months
  A complete blood cell differential will be taken, including neutrophilia and eosinophilia.
Serum Club cell secretory protein | Baseline (day 0)
Serum Club cell secretory protein | 12 months
Sputum bacteriology | Baseline (day 0)
Sputum bacteriology | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jérémy Charriot, MD, Study Director — University Hospital, Montpellier
Locations (3):
- France (3):
  - University Hospitals of Bordeaux, Bordeaux
  - University Hospitals of Montpellier, Montpellier
  - University Hospitals of Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: Yes
The general goal is to make the study data available to interested researchers as well as to provide proof of transparency for the study. Data (and an accompanying data dictionary) will be de-identified and potentially further cleaned or aggregated as the investigators deem necessary to protect participant anonymity.
  Data will be made available to persons who address a reasonable request to the study director and fulfil the requirements stipulated by the French CNIL (Commission Nationale de l'Informatique et des Libertés : https://www.cnil.fr/professionnel).
Time Frame: As close to "real time" as possible, the following supporting information will be made public:
  * Study Protocol (to be published in an appropriate journal).
  * Statistical Analysis Plan
  * Participant Information materials
  * Analytic code
  These will be posted and registered on osf.io and/or clinicaltrials.gov (if not published).
  Datasets can be requested after the publication process has been completed.
Access Criteria: The conditions under which members of the public will be granted access to datasets are:
  * The data will be used/examined in a not-for-profit manner;
  * The data will not be used in an attempt to identify a participant or group of participants;
  * The user does not work for a private insurance company;
  * The data will not be used in support of any kind of private insurance policy or health penalties;
  * The data will be used/examined for the advancement of science/teaching while respecting participant/patient privacy and rights;
  * The user will state why they wish to access the data.
  * The appropriate CNIL approval has been obtained by the user.
URL: https://osf.io/kr5pa/